CLINICAL TRIAL: NCT07312617
Title: Comparison of Anatomical and Subjective Short-term Outcomes of TOT, TVT, and Burch Colposuspension: A Randomized Controlled Trial Using Transperineal Ultrasound
Brief Title: Short-Term Outcomes of TOT, TVT, and Burch Surgery Assessed by Transperineal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, gizem boz izceyhan, doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37/2023
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Stress Urinary Incontinence in Women; Pelvic Floor Disorders
Keywords: sui; tpus
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Suburethral Slings

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of three parallel intervention groups (TOT, TVT, or Burch colposuspension), and each participant received only one type of surgical intervention. Outcomes were assessed and compared between groups during the same follow-up period.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tot (Active Comparator): Participants underwent mid-urethral sling surgery for the treatment of stress urinary incontinence.
  Interventions: Procedure: Transobturator Tape (TOT) Procedure
- tvt (Active Comparator): Participants in this arm underwent tension-free vaginal tape (TVT) surgery for the treatment of stress urinary incontinence.
  Interventions: Procedure: Tension-Free Vaginal Tape (TVT) Procedure
- Burch Colposuspension (Active Comparator): Participants in this arm underwent Burch colposuspension surgery for the treatment of stress urinary incontinence.
  Interventions: Procedure: Burch Colposuspension Procedure

INTERVENTIONS:
Procedure: Transobturator Tape (TOT) Procedure — Placement of a synthetic tape beneath the mid-urethra via the transobturator route.
  Other Names: tot
  Arms: tot
Procedure: Tension-Free Vaginal Tape (TVT) Procedure — Placement of a synthetic tape beneath the mid-urethra using a retropubic approach.
  Arms: tvt
Procedure: Burch Colposuspension Procedure — Suspension of the anterior vaginal wall to the iliopectineal (Cooper's) ligament using non-absorbable sutures.
  Arms: Burch Colposuspension

SUMMARY:
Stress urinary incontinence is a common condition in women and is often treated with surgical procedures such as transobturator tape (TOT), tension-free vaginal tape (TVT), and Burch colposuspension. Although these procedures are widely used, there is limited information comparing their short-term anatomical and patient-reported outcomes using imaging techniques.

The aim of this study is to compare the short-term anatomical and subjective outcomes of TOT, TVT, and Burch colposuspension in women with stress urinary incontinence. Transperineal ultrasonography will be used to assess anatomical changes before surgery and during follow-up. Patient-reported outcomes and clinical findings will also be evaluated.

The results of this study may help improve the understanding of surgical outcomes in stress urinary incontinence and support clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older
* Diagnosis of stress urinary incontinence based on clinical evaluation
* Candidates for surgical treatment with transobturator tape (TOT), tension-free vaginal tape (TVT), or Burch colposuspension
* Ability to provide written informed consent
* Willingness to participate in the study and comply with follow-up visits

Exclusion Criteria:

* Mixed or urge-predominant urinary incontinence
* Previous anti-incontinence or pelvic floor surgery
* Neurogenic bladder disorders
* Active urinary tract infection at the time of evaluation
* Pregnancy or planned pregnancy during the study period
* Known pelvic malignancy
* Inability to undergo transperineal ultrasonographic evaluation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Urethrovesical and Urethral Angles Assessed by Transperineal Ultrasound | Baseline (preoperative) and 3 months postoperatively
  The primary outcome is the change in urethrovesical and urethral angles measured by transperineal ultrasonography before surgery and at 3 months after surgery.

SECONDARY OUTCOMES:
Subjective Improvement in Stress Urinary Incontinence Symptoms | Baseline and 3 months postoperatively
  Subjective outcomes were assessed using the Urogenital Distress Inventory-Short Form (UDI-6) and the Incontinence Impact Questionnaire-Short Form (IIQ-7). For both scales, scores range from 0 to 100, where higher scores indicate a greater impact of symptoms and worse quality of life.

OTHER OUTCOMES:
Comparison of Anatomical Outcomes Between Surgical Techniques | 3 months postoperatively
  Anatomical outcomes assessed by transperineal ultrasonography were compared between the TOT, TVT, and Burch colposuspension groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women and Children Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No